CLINICAL TRIAL: NCT00533247
Title: Preemptive Anti-Inflammatory Use of Celecoxib in Knee Arthroplasty Surgery: a Double Blinded, Placebo-Controlled Study.
Brief Title: Arthroplasty Inflammation Prophylaxis With Celecoxib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zanbilowicz, Adam, DPM MS (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAC01
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Postoperative Pain
Keywords: Cox-2 Inhibitor; Pre-emptive Pain; Preoperative Pain; Pain Prophylaxis; Celebrex; Celecoxib
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
This double blinded, placebo controlled, study seeks to determine the efficacy of preoperative anti-inflammatory therapy on the reduction of postoperative pain in knee arthroplasty surgery. Pre-emptive use of NSAIDS has demonstrated only modest reduction in post-operative pain in previous studies. However, the short duration of dosing in those studies did not capitalized on the anti-inflammatory properties of NSAIDS. Short-term use of NSAIDS only provides pain relief and does not address inflammation. Traditional NSAIDS cannot be used preoperatively due to platelet effects. Celecoxib, however, is both an analgesic and anti-inflammatory, but does not interfere with bleeding. It can therefore be safely used before surgery. This study hypothesizes that the use of celecoxib for seven days preoperatively reduces postoperative inflammation and consequently pain. A detailed Medline search has not identified any studies into the preoperative use of an NSAID at a dosing level that achieves anti-inflammatory effects.If effective in reducing postoperative pain, this research could lead to a new understanding of the role inflammation plays in orthopedic procedures and other elective procedures and thus improve patient outcomes in the future.

DETAILED DESCRIPTION:
Abstract:

This double blinded, placebo controlled, study seeks to determine the efficacy of preoperative anti-inflammatory therapy on the reduction of postoperative pain in knee arthroplasty surgery. Pre-emptive use of NSAIDS has demonstrated only modest reduction in post-operative pain in previous studies. However, the short duration of dosing in those studies did not capitalized on the anti-inflammatory properties of NSAIDS. Short-term use of NSAIDS only provides pain relief and does not address inflammation. Traditional NSAIDS cannot be used preoperatively due to platelet effects. Celecoxib, however, is both an analgesic and anti-inflammatory, but does not interfere with bleeding. It can therefore be safely used before surgery. This study hypothesizes that the use of celecoxib for seven days preoperatively reduces postoperative inflammation and consequently pain. A detailed Medline search has not identified any studies into the preoperative use of an NSAID at a dosing level that achieves anti-inflammatory effects.If effective in reducing postoperative pain, this research could lead to a new understanding of the role inflammation plays in orthopedic procedures and other elective procedures and thus improve patient outcomes in the future.

Purpose and Significance:

It is commonly accepted that inflammation significantly increases pain. To date, no study has examined the potential benefits of preemptively treating inflammation before surgery. While the analgesic effects of NSAIDs have a rapid onset, the maximal anti-inflammatory effect can take one to three weeks to be realized. Due to bleeding concerns, traditional NSAIDS such as naprosyn or ibuprofen cannot, and have not, been used preoperatively. Following surgery, the inflammatory cascade of cells and chemical mediators inundates the surgical wound and creates acute inflammation. Once this has happened NSAIDs have missed the opportunity to treat this acute inflammation. Post-operative and single dose preoperative use of NSAIDs act exclusively as analgesics. Since celecoxib has no impact on postoperative bleeding, it can be safely administered preoperatively. With adequate time before an elective operation, one has the opportunity to reach steady state pharmacokinetics and a sufficient serum level to prevent inflammation -- and therefore pain

Aims of Study:

1. Compare the efficacy of a seven-day preoperative course of celecoxib 200mg taken orally once daily against the efficacy of a single preoperative 200mg dose administered on the day of the operation in reducing postoperative pain.

Endpoints:

Primary Endpoint: Comparison of the total pain rating in group receiving seven days of preoperative of celecoxib against total pain rating in the group receiving the single dose of celecoxib. Total Pain will be calculated by summing ten point verbal rating scale (VRS) at time intervals of: "When you woke up following surgery," 24 hours postoperatively and 48 hours postoperatively.

Additional endpoints:

1. Comparison of pain rating VRS "When you woke up following surgery," and at 24 hours and 48 hours postoperatively in the two study groups
2. Comparison of patient reported maximum pain on VRS in the study groups.

Methods:

Study Size

50 Patients undergoing total knee arthroplasty will receive celecoxib 200mg once daily for seven days preoperatively 50 Patients undergoing total knee arthroplasty will receive placebo once daily for six days preoperatively and on the day of the operation will receive a single dose of celecoxib 200mg.

In order to be able to detect a difference of 2 points on the 0-10 scale between either intervention group and placebo group, with 80% power (at 5% 2 sided significance level and assuming a SD of 3.5) 50 subjects per group would be sufficient. That detectible difference combined with the assumed SD is equivalent to a moderate to large effect size (i.e. one that is clinically relevant).

Selection and Recruitment of Participants

Consecutive patients scheduled for knee arthroplasty surgery who meet the study inclusion criteria would be enrolled and randomized to either the seven day course group or the single dose/placebo group. Randomization will be done via sealed, coded study packages that include either medication or placebo. These packages will be dispensed to the patients

Physicians recruiting patients will will dispense study information brochures. If patients are interested in participating, the study nurse will then contact them and she will provide full study details and obtain informed consent.

Exclusion Criteria - Subjects will be excluded from the study for the following reasons:

* Allergy to non-steroidal anti-inflammatory medications
* Subjects must not be taking another NSAID while the study is conducted
* Bleeding disorder
* Impaired renal function (serum creatinine >1.2 x upper limit of normal)
* Liver Disease (SGPT(ALT) or SGOT(AST) > 1.5x upper limit of normal)
* Heart Disease
* Ulcers
* Taking an ACE inhibitor
* Taking a diuretic
* Must not be taking an NSAID on a daily basis during the study period
* Pregnant or planning to start a pregnancy soon

Medication Dose

Celecoxib begins to act as an analgesic within minutes of oral administration. Anti-inflammatory efficacy of NSAIDS has been shown to have a latency of one to two weeks. Ibuprofen, for example requires a dosing of 1200mg/day (the maximum over the counter dose) and reaches peak anti-inflammatory efficacy in 7-14 days. For other NSAIDS, anti-inflammatory dosing is at a higher level than at analgesic dosing. Celecoxib reaches steady state in five days. To ensure that this study achieves steady state levels of celecoxib in the serum, and that it is acting as an anti-inflammatory rather than just as an analgesic a one to two-week time frame is needed. To improve patient compliance, once daily dosing of 200mg was selected over twice daily.

Pain Assessment

Pain assessments will be made on prepared pain forms that contain a visual pain scale. Data will be collected by patients on their pain diary and will be reported to the researchers via a toll-free phone number. The study nurse will also contact patients directly at each study interval to ensure collection of data.

Data Collection

Data collection will be done by telephone conversation with patients once they have returned home from the surgery as they recover. Patients will be asked to report their pain on a ten-point scale. The scale will be described to the patient as "zero being no pain and ten being the worst pain imaginable."

Patients will have diaries dispensed and will be asked to telephone a toll free number at the appropriate times. Additionally, the study nurse will call patients at the study data collection intervals (i.e "When you woke up following surgery," 24 hours and 48 hours) to ensure data collection. Patients will also be asked to state the number indicating the worst pain that they experienced during their postoperative period - this will be asked/recorded at the 48 hour postoperative interval.

Statistical Analysis

Study data will be analyzed by an independent statistician.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients undergoing knee arthroplasty

Exclusion Criteria:

Subjects will be excluded from the study for the following reasons:

* Allergy to non-steroidal anti-inflammatory medications
* Subjects must not be taking another NSAID while the study is conducted
* Bleeding disorder
* Impaired renal function (serum creatinine >1.2 x upper limit of normal)
* Liver Disease (SGPT(ALT) or SGOT(AST) > 1.5x upper limit of normal)
* Heart Disease
* Ulcers
* Taking an ACE inhibitor
* Taking a diuretic
* Must not be taking an NSAID on a daily basis during the study period
* Pregnant or planning to start a pregnancy soon

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Compare total pain rating in group receiving 7day celecoxib against in 1 dose celecoxib

SECONDARY OUTCOMES:
1. Comparison of pain rating VRS "When you woke up following surgery," and at 24 hours and 48 hours postoperatively in the two study groups
Comparison of patient reported maximum pain on VRS in the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Zanbilowicz, BA DPM MS, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver, British Columbia, Canada